CLINICAL TRIAL: NCT01243411
Title: A Phase 3, Open-label Study of the Safety and Effectiveness of AA4500 Administered Twice Per Treatment Cycle for up to Four Treatment Cycles (2 x 4) in Men With Peyronie's Disease
Brief Title: A Study of AA4500 in Men With Peyronie's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-802
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's Disease, penile plaque, penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 (Experimental): collagenase clostridium histolyticum
  Interventions: Biological: AA4500

INTERVENTIONS:
Biological: AA4500 — 2 injections separated by at least 24 hours but not more than 72 hours, repeated after 42 days (± 5 days) for up to 4 treatment cycles (ie, total of up to 8 injections per subject)
  Other Names: XIAFLEX

SUMMARY:
This study is a Phase 3, open-label study of the safety and efficacy of AA4500 0.58 mg in subjects with Peyronie's disease. Subjects will be screened for study eligibility within 21 days before the initial injection of study drug in the first treatment cycle.

After up to four treatment cycles, each subject will be followed for additional safety and efficacy assessments on Days 168 (± 7 days) and 252 (± 7 days) (nominal weeks 24 and 36).

After the final injection of each treatment cycle, the investigator will model the plaque in an attempt to stretch or elongate the plaque. If the subject's penile curvature is reduced to <15° after the first, second, or third cycle of injections or if the investigator determines further treatment is not clinically indicated (eg, adverse events; allergic reaction), subsequent treatment cycles will not be administered.

Approximately 300 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

No subject should be enrolled until all eligibility criteria have been satisfied. Subjects who receive placebo in a previous Auxilium-sponsored study may enroll in this study provided they continue to meet the eligibility requirements. To qualify for the study a subject must:

1. Be a male and be ≥ 18 years of age
2. Be in a stable relationship with a female partner/spouse for at least 3 months before screening and be willing to have vaginal intercourse with that partner/spouse
3. Have symptom(s) of Peyronie's disease for at least 12 months before the first dose of study drug and have evidence of stable disease as determined by the investigator
4. Have penile curvature of at least 30° in the dorsal, lateral, or dorsal/lateral plane at screening. It must be possible to delineate the single plane of maximal curvature for evaluation during the study
5. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile
6. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
7. Be able to read, complete and understand the various rating instruments in English or the appropriate local language for the country in which the study is being performed.

   -

Exclusion Criteria:

A subject will be excluded from study participation if he:

1. Has a penile curvature of less than 30° or greater than 90° at the screening visit
2. Has any of the following conditions:

   * Chordee in the presence or absence of hypospadias
   * Thrombosis of the dorsal penile artery and/or vein
   * Infiltration by a benign or malignant mass resulting in penile curvature
   * Infiltration by an infectious agent, such as lymphogranuloma venereum
   * Ventral curvature from any cause
   * Presence of an active sexually transmitted disease
   * Known active hepatitis B or C
   * Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
3. Has previously undergone surgery for Peyronie's disease
4. Fails to have an erection which in the opinion of the investigator is sufficient to accurately measure the subject's penile deformity after administration of prostaglandin E1 or trimix
5. Has a calcified plaque as evident by appropriate radiographic evaluation, penile x-ray or penile ultrasound that would prevent proper injection of study medication (penile ultrasound only in EU countries). Non-contiguous stippling of calcium is acceptable for inclusion provided the calcium deposit does not interfere with the injection of AA4500 into the plaque
6. Has an isolated hourglass deformity of the penis
7. Has the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of the local anesthetic would interfere with the injection of AA4500 into the plaque
8. Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
9. Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [> 500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, pentoxifylline, over-the-counter erectile dysfunction medications, or steroidal anti-inflammatory drugs) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
10. Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6-month period before screening or plans to have ESWT at any time during the study
11. Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
12. Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
13. Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
14. Has a penile Duplex Doppler ultrasound evaluation at screening that shows compromised penile hemodynamics that in the opinion of the investigator is clinically significant
15. Has uncontrolled hypertension, as determined by the investigator
16. Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
17. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits
18. Has received an investigational drug or treatment within 30 days before the first dose of study drug, except for subjects who receive one treatment cycle of AA4500 in Study AUX-CC-805
19. Has a known systemic allergy to collagenase or any other excipient of AA4500
20. Has a known allergy to any concomitant medication required as per the protocol
21. Has received anticoagulant medication (except for ≤ 165 mg aspirin daily or ≤ 800 mg of over-the-counter NSAIDS daily) during the 7 days before each dose of study drug
22. Has received any collagenase treatments within 30 days of the first dose of study drug, except for subjects who receive one treatment cycle of AA4500 in Study AUX-CC-805
23. Has, at any time, received AA4500 for the treatment of Peyronie's disease, except for subjects who receive one treatment cycle of AA4500 in Study AUX-CC-805

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J. Kaufman, MD, Study Director — Auxilium Pharmaceuticals, Inc.
Locations (39):
- United States (13):
  - Urology Associates Medical Group, Burbank, California
  - Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - The Urology Center, P.C., New Haven, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Urology Specialists, S.C., Chicago, Illinois
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Metropolitan Urology, P.S.C., Jeffersonville, Indiana
  - Maimonides Medical Center, Division of Urology, Brooklyn, New York
  - University Urology Associates, New York, New York
  - Tristate Urologic Services PSC, Inc./ dba TUG Research, Cincinnati, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology of Virginia-Sentara Medical Group, Norfolk, Virginia
  - Virginia Urology, Richmond, Virginia
- Denmark (4):
  - Aarhus Universitiy Hospital, Aalborg Sygehus, Aalborg
  - Frederiksberg Hospital, Frederiksberg
  - Frederikssunds Hospital, Frederikssund
  - Klinik for seksuelle dysfunktioner, Gentofte Municipality
- France (2):
  - Centre Hospitalier Edouar Herriot, Lyon
  - Hopital Henri Gabrielle, Saint-Genis-Laval
- Germany (5):
  - Universitatsklinikum Freiburg, Abteilung Urologie, Freiburg im Breisgau
  - Private Practice of Urology/Andrology, Hamburg
  - Uro-Onkologische Praxis Dr. von Keitz, Marburg
  - Urologische Gemeinschaftspraxis Reutlingen, Reutlingen
  - Universitatsklinikum Tubingen, Tübingen
- Italy (2):
  - University of Naples "Federico II", Naples
  - Universitiy Tor Vergatat of Rome, Rome
- New Zealand (6):
  - Waitemata Urology Research North Shore Hospital, Takapuna, Auckland
  - Tauranga Urology Research Ltd., Tauranga, Bay of Plenty
  - Primorus Clinical Trials Ltd., Christchurch, Canterbury
  - CURT Medical Trials Trust Board Inc., Christchurch, Canterbury
  - Cardinal Points Research Ltd., Whangarei, Northland
  - Wellington Urology Associates, Wellington South, Wellington Region
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital La Zarzuela, Madrid
- Sweden (3):
  - Specialistmottagningen i urologi, Gothenburg
  - Carlshamns Specialistklinik, Karlshamn
  - Akademiska Sjukhuse, Uppsala
- United Kingdom (2):
  - St. Peter's Andrology Centre, London
  - Sunderland Royal Hospital, Sunderland

REFERENCES:
- [Derived] Levine LA, Cuzin B, Mark S, Gelbard MK, Jones NA, Liu G, Kaufman GJ, Tursi JP, Ralph DJ. Clinical safety and effectiveness of collagenase clostridium histolyticum injection in patients with Peyronie's disease: a phase 3 open-label study. J Sex Med. 2015 Jan;12(1):248-58. doi: 10.1111/jsm.12731. Epub 2014 Nov 12. PMID 25388099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Includes all subjects who were enrolled and received at least 1 dose of study drug; subjects who were enrolled but not treated were excluded from the population
Period: Overall Study
Arm/Group | AA4500
Started | 347
Completed | 306
Not Completed | 41
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 10
Not completed — Adverse Event | 5
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | AA4500
Number analyzed (Participants) | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 289
  >=65 years | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 347
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 325
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 333
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  France | 13
  United States | 102
  Spain | 21
  Denmark | 42
  Germany | 41
  Italy | 24
  United Kingdom | 17
  New Zealand | 54
  Sweden | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Penile Curvature
Description: A negative value in the percentage change from baseline in penile curvature deformity (angle measured in degrees) indicates less curvature.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the modified intent-to-treat (mITT) population.
Measure: Mean (Standard Deviation); unit: percentage of curvature change
Arm/Group | AA4500
Number analyzed (Participants) | 238
percentage of curvature change | -34.4 (25.21)

2. Primary Outcome: Change From Baseline in the Peyronie's Disease Bother Domain of the Peyronie's Disease Questionnaire (PDQ)
Description: Peyronie's disease bother score range 0 (no issue or not at all bothered) to 4 (extremely bothered) on 4 questions; total score range 0 to 16. A decrease in the change from baseline total score in the Peyronie's disease bother domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 238
units on a scale | -3.3 (3.46)

3. Secondary Outcome: Change From Baseline in the Severity of Peyronie's Disease Symptoms Domain of the PDQ
Description: Peyronie's disease symptoms (physical and psychological) severity score range 0 (none) to 4 (very severe) on 6 questions; total score range 0 to 24. A decrease in the change from baseline total score in the Peyronie's disease symptoms domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 238
units on a scale | -4.2 (5.14)

4. Secondary Outcome: Change From Baseline in the Penile Pain Domain of the PDQ in Subjects With Baseline Penile Pain Score ≥4
Description: Penile pain scale range 0 (no pain) to 10 (extreme pain) on 3 questions; total score range 0 to 30. A decrease in the change from baseline total score in the penile pain domain of the PDQ is indicated by a negative number. Subjects were required to have a penile pain score of 4 or greater at baseline.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population; this population only includes those subjects in the mITT population with a baseline penile pain score of 4 or greater.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 114
units on a scale | -5.3 (4.93)

5. Secondary Outcome: A Responder Analysis Based on Subject Overall Global Assessment
Description: Subject overall global assessment of Peyronie's disease score range -3 (much worse) to 3 (much improved). A score of 1 (improved in a small but important way), 2 (moderately improved), or 3 indicate a responder.
Time Frame: Week 36
Population: Efficacy is based on the mITT population.
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 238
participants
  Responder Status - Yes | 172
  Responder Status - No | 66

6. Secondary Outcome: Change in the Overall Satisfaction Domain of the International Index of Erectile Function (IIEF)
Description: Overall satisfaction domain of the IIEF score range 0 to 5 on 2 questions where higher scores indicate improved function or satisfaction; total score range 0 to 10.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 238
units on a scale | 1.1 (2.23)

7. Secondary Outcome: Change From Baseline in Penile Plaque Consistency
Description: Penile plaque consistency score range 1 (non-palpable) to 5 (hard). A decrease in the change from baseline in penile plaque consistency is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 238
units on a scale | -0.8 (0.93)

8. Secondary Outcome: A Composite Responder Analysis Based on Change From Baseline in Penile Curvature and in the Peyronie's Disease Bother Score
Description: A composite responder is indicated by
  * a percent reduction from baseline in penile curvature greater than or equal to the threshold, and
  * a reduction from baseline in Peyronie's disease bother score greater than or equal to the threshold, or change in the overall sexual activity within the last 3 months to having vaginal intercourse from no vaginal intercourse at screening.
Time Frame: Week 36
Population: Composite responder analysis is based on the intent-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 347
participants
  Responder - Yes | 177
  Responder - No | 140
  Responder - Missing | 30

9. Secondary Outcome: Change From Baseline in Penile Length
Description: A negative value represents a reduction in measurement from baseline.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | AA4500
Number analyzed (Participants) | 238
centimeters | 0.4 (1.11)

ADVERSE EVENTS:
Arm/Group | AA4500
Serious Adverse Events (participants affected / at risk) | 13/347
Other Adverse Events (participants affected / at risk) | 297/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AA4500 (N=347)
Penile haematoma (Reproductive system and breast disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Deep vein thrombosis (Vascular disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Device occlusion (General disorders) | 1 — Right coronary artery in-stent occlusion
Fracture of penis (Injury, poisoning and procedural complications) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Mania (Psychiatric disorders) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=347)
Penile haematoma (Reproductive system and breast disorders) | 178 (356)
Penile pain (Reproductive system and breast disorders) | 120 (261)
Injection site pain (General disorders) | 93 (171)
Penile swelling (Reproductive system and breast disorders) | 91 (138)
Injection site haematoma (General disorders) | 84 (139)
Penile haemorrhage (Reproductive system and breast disorders) | 79 (203) — penile ecchymosis
Penile oedema (Reproductive system and breast disorders) | 49 (120)
Injection site swelling (General disorders) | 40 (68)
Painful erection (Reproductive system and breast disorders) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other